CLINICAL TRIAL: NCT00653601
Title: Bridging Therapy in Patients at High Risk for Stent Thrombosis Undergoing Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Dr Sanjay Kaul, PI, CSMC
Other Study IDs: Pro00014008
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Bleeding; Thrombosis
Keywords: GPI; glycoprotein IIb/IIIa inhibitor; Aggrastat; Tirofiban; Verify now; platelet function testing; bridge therapy
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 mL of blood for testing X 5 per patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients who receive bridge therapy with tirofiban who were previously on plavix for drug eluting or bare metal stent prior to scheduled invasive procedures
- 2: Patients who do NOT receive bridge therapy previously on plavix for drug eluting or bare metal stent prior to scheduled invasive procedures. This will entail of a matching case-control for the following characteristics.
  * # of RF for stent thrombosis
  * types of stents
  * time frame when the stents were placed
  * procedure type

SUMMARY:
Patients who have undergone placement of coronary stents require dual antiplatelet therapy with Plavix and aspirin to prevent the serious complication of in-stent thrombosis. Some of these patients will require surgery while on dual antiplatelet therapy. This poses a challenge because being on Plavix is associated with higher risks of perioperative bleeding, but stopping Plavix puts patients at increased risk for in-stent thrombosis.

Currently, the ACC/AHA guidelines recommend discontinuation of Plavix five days prior to surgery to prevent bleeding complications. However, there are no universal recommendations for preventing in-stent thrombosis. Some experts recommend the use glycoprotein IIb/IIIa inhibitors (short-acting antiplatelet agents) as "bridging therapy" during the high-risk perioperative period. Although these agents should be beneficial based on theory, there is currently no published data on their effectiveness for this purpose.

The current study proposes to evaluate the value of Aggrastat (a short-acting intravenous platelet glycoprotein IIb/IIIa inhibitor) in decreasing the risk of in-stent thrombosis without increasing the risk of perioperative bleeding.

DETAILED DESCRIPTION:
A. D/C clopidogrel 5 days prior to surgery

B. Continue ASA (Increase dose to 325 mg until prohibitive bleeding risk)

C. Check baseline IIb/IIIa and P2Y12 via the Verify Now device prior to initiating tirofiban

D. Start Tirofiban 2 days prior to the procedure (Patient MUST be on a monitored bed)

* Load Tirofiban ONLY if P2Y12 (Verify Now Assay) platelet inhibition is < 20% OTHERWISE initiate only the continuous infusion dose
* Creatinine clearance > 30mL/min: Tirofiban 0.4 mcg/kg/min for 30 minutes, followed by continuous infusion at 0.1 mcg/kg/min
* Creatinine clearance < 30mL/min: Tirofiban 0.2 mcg/kg/min for 30 minutes, followed by continuous infusion of 0.05 mcg/kg/min

E. Check steady state IIb/IIIa inhibitor verify now assay (>8 hour after initiation)

F. Hold Tirofiban 12 hours prior to procedure

G. Check IIb/IIIa inhibitor verify now assay (10-12 hours after Tirofiban is discontinued)

H. CBC pre and post op

I. Reload clopidogrel> 24 hours post op (300 mg X 1 then 75 mg daily) unless prohibitive bleeding risk

J. Reduce ASA to pre-procedure dose. Restart ASA, 24 hours port-op if it was D/C prior to procedure

K. Check P2Y12 via the Verify Now device post-loading dose of clopidogrel (test cannot be performed w/in 48 hours of the D/C of IIb/IIIa inhibitor (tirofiban)

ELIGIBILITY:
Inclusion Criteria:

* Patients' with BMS/DES on plavix prior to surgery who are in need of an elective procedures

Exclusion Criteria:

* Patients' with BMS/DES on NOT plavix prior to surgery who are in need of an elective procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' with BMS/DES on plavix prior to surgery who are in need of an elective procedures
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
In-stent thrombosis as assessed by acute coronary syndromes of unstable angina/non-ST elevation myocardial infarction or ST-elevation myocardial infarction during the hospitalization. | until discharge

SECONDARY OUTCOMES:
Platelet function using the Verify Now device: T1 - at admission (2-3 days after the D/C of Plavix and prior to initiation of Aggrastat infusion); T2 - > 8 hours after initiation of Aggrastat; T3 - pre-operative; T4 - post loading dose of clopidogrel. | until discharge
Bleeding as assessed by hematocrit values obtained immediately pre-operative, immediately post-operative, and prior to discharge In addition, the use of blood products (pRBCs, platelets, FFP) will be assessed. | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kaul, MD, Principal Investigator — Attending physician
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States